CLINICAL TRIAL: NCT00923936
Title: Pilot Study of Liposomal Doxorubicin Combined With Bevacizumab Followed by Bevacizumab Monotherapy in Adults With Advanced Kaposi s Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Robert Yarchoan, Branch Chief HIV and AIDS Malignancy Branch, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 090130; 09-C-0130; NCT00902239 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Results first posted 2017-06-16 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-06

CONDITIONS: Sarcoma, Kaposi
Keywords: Kaposi's Sarcoma; HIV; Doxil; VEGF; Bevacizumab
MeSH Terms: conditions — Sarcoma, Kaposi | interventions — liposomal doxorubicin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- KS;classic/HIV+not improved on antiviral (Active Comparator): Kaposi's Sarcoma (KS) in patients who are Human immunodeficiency virus (HIV) Negative, HIV infected with stable disease for one year despite antiretroviral therapy or progressive disease despite 4 months of antiretroviral therapy.
  Interventions: Drug: Liposomal Doxorubicin; Drug: Bevacizumab
- All other advanced HIV-asociated KS (Active Comparator): All other patients with advanced acquired immune deficiency syndrome (AIDS)-associated KS
  Interventions: Drug: Liposomal Doxorubicin; Drug: Bevacizumab

INTERVENTIONS:
Drug: Liposomal Doxorubicin — Induction phase dose: Intravenous (IV) bevacizumab 15 mg/kg once, followed 7 days later by liposomal doxorubicin mg/m^2 and bevacizumab every 3 weeks for six cycles.
  Other Names: Doxil
Drug: Bevacizumab — Induction phase dose: Intravenous (IV) bevacizumab 15 mg/kg once, followed 7 days later by liposomal doxorubicin mg/m^2 and bevacizumab every 3 weeks for six cycles. Maintenance phase dose: IV bevacizumab every 3 weeks for 11 cycles.
  Other Names: Avastin

SUMMARY:
Background:

* The drug liposomal doxorubicin is approved by the U.S. Food and Drug Administration (FDA) for the treatment of Kaposi's sarcoma (KS). A second drug, bevacizumab, is a biologic agent (such as antibodies, interleukins, and vaccines) that stops abnormal blood supply to tumors. Bevacizumab is approved by the FDA, in combination with other drugs, for the treatment of breast cancer, colon cancer, and lung cancer.
* Researchers are now studying the combination of liposomal doxorubicin with bevacizumab as a novel approach to the treatment of advanced KS. Researches will be measuring KS tumor responses to this combination to determine whether the drugs might have anti-KS activity.

Objectives:

* To estimate the overall response rate (ORR) of six cycles of liposomal doxorubicin combined with bevacizumab in patients with advanced KS.
* To evaluate the safety of the regimen and to estimate the complete response rate after six cycles, the median number of cycles needed to obtain a partial response, and the 12-month progression-free survival.

Eligibility:

* Patients 18 years or older with relatively severe acquired immune deficiency syndrome (AIDS)-related KS or patients with KS unrelated to AIDS or human immunodeficiency virus (HIV) infection, whose KS that can be evaluated for potential response to therapy and meet a number of other criteria.
* Women who are pregnant or breastfeeding are not eligible.
* Other ineligibility criteria include surgery within 4 weeks, chemotherapy within 3 weeks, heart disease, hemoptysis (coughing up blood), or gastrointestinal bleeding.

Design:

* Researchers will conduct the following tests before the start of the study:
* Physical examination and a detailed medical history.
* A biopsy.
* Blood and urine tests.
* Treatment will include two phases, an induction phase and a maintenance phase:
* Induction phase dose: Intravenous (IV) bevacizumab 15 mg/kg once, followed 7 days later by liposomal doxorubicin mg/m2 and bevacizumab every 3 weeks for six cycles.

Maintenance phase dose: IV bevacizumab every 3 weeks for 11 cycles.

* Monitoring will include a review of side effects, physical exam (including blood pressure), and blood and urine samples; following the induction phase, the patient will receive a multi gated acquisition scan and electrocardiography (EKG) to record electrical activity in the heart.
* Research tests include blood and saliva samples, additional biopsies (optional), and noninvasive imaging.
* Treatment is stopped if any of the following occur: completion of 1 year of therapy, progressive KS, patient preference, or unacceptable toxicity.
* Post-treatment evaluations include clinic visits every 3 months or as needed up to 2 years, and blood and saliva samples (for research).

DETAILED DESCRIPTION:
Background:

* Standard treatment for advanced Kaposi's sarcoma (KS) is a liposomal anthracycline, plus antiretroviral therapy (HAART) in patients with human immunodeficiency virus (HIV).
* KS is not curable and relapses are common. Prolonged use of liposomal anthracyclines with cumulative dosing exceeding 550 mg/m(2) is frequently required.
* KS is notable for pathogenic autocrine and paracrine vascular endothelial growth factor (VEGF) signaling. The monoclonal antibody, bevacizumab is a rational agent for the treatment of KS.
* Preliminary results from our phase II study of bevacizumab monotherapy, 03-C0110, suggest that bevacizumab has promising activity in the treatment of KS.
* The combination of anti-angiogenic therapy with cytotoxic chemotherapy has been a successful strategy in KS as well as other solid tumors.
* This pilot study will evaluate the activity and safety of liposomal doxorubicin combined with bevacizumab followed by bevacizumab maintenance in patients with advanced KS. A goal of this combination strategy is to develop a tolerable and highly active regimen that would limit the need for prolonged anthracycline use.

Objectives:

* The primary objective is to estimate the overall response rate (ORR) of six cycles of liposomal doxorubicin combined with bevacizumab in patients with advanced KS.
* Secondary objectives include evaluation of the safety of the regimen, as well as estimation of the complete response rate after 6 cycles, the median number of cycles need to obtain a partial response, and 12-month progression-free survival.

Eligibility:

Inclusion criteria:

* Age greater than or equal to 18
* Biopsy proven KS
* Indication for chemotherapy
* Any HIV status
* Normal multigated acquisition scan (MUGA)
* Able to tolerate aspirin 81 mg
* systolic blood pressure (SBP) <150, diastolic blood pressure (DBP) <90
* Urine protein <1+ or 500mg/24hrs

Exclusion Criteria:

* Surgery within 4 weeks
* Thrombo-embolic disease
* Chemotherapy within 3 weeks
* Hemoptysis or severe gastrointestinal bleeding, unless caused by KS
* Pregnancy or breast feeding

Design:

* This is an open label, single center pilot with 2 cohorts. Cohort 1: HIV negative, HIV infected with stable KS despite 1 year of HAART with HIV viremic control, or HIV infected with progressive KS despite 4 months of HAART with HIV viremic control. Cohort 2: All other patients with advanced AIDS-associated KS.
* Subjects will receive bevacizumab 15 mg/kg and liposomal doxorubicin 20 mg/m(2) every 3 weeks until complete response (CR) or a maximum of 6 cycles. Those with stable disease or better will continue on bevacizumab 15 mg/kg monotherapy every 3 weeks for 11 cycles. HIV infected subjects will receive HAART.
* ORR will be calculated with 80% CI for each cohort separately. If estimates in the two cohorts are similar (p>0.30 by a Fisher s exact test), they may be combined to form a somewhat more precise estimate of ORR after 6 cycles of treatment.
* A total of 10 evaluable patients will be accrued in each cohort.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Age greater than or equal to 18 years
2. Kaposi s sarcoma pathologically confirmed by Center for Cancer Research (CCR) pathology
3. Evaluable Kaposi's sarcoma (KS) involving the skin and/or viscera, including at least one of the following:

   * KS of the skin with greater than or equal to 5 KS lesions that are evaluable by non-invasive methods that have not been treated with local therapeutic modalities
   * Pulmonary KS evaluable by computed tomography (CT) scan
   * Gastrointestinal KS evaluable by direct visualization or fiberoptic instrumentation
   * Biopsy proven lymph node involvement measurable by CT scan
4. Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
5. Life expectancy > 6 months
6. At least one of the following indications for therapy:

   * Pulmonary involvement
   * Visceral involvement
   * Pain
   * Edema
   * Substantial lymph node involvement
   * Ulcerating lesions
   * Decreased range of joint motion due to KS
   * Multiple lesions not amenable to local therapy
   * Significant psychological impact leading to social withdrawal
7. Patients with human immunodeficiency virus (HIV) infection must be willing to comply with a regimen of highly active antiretroviral therapy (HAART).
8. Patients may have received any number of prior therapies, including monotherapy with liposomal doxorubicin or bevacizumab
9. Blood pressure

   * Systolic blood pressure (SBP) < 150 mm/Hg
   * Diastolic blood pressure (DBP) < 90 mm/Hg
   * Patients receiving anti-hypertensive medicines must be on a stable regimen for at least 1 month
10. Ejection fraction (EF) > 50% by multigated acquisition scan (MUGA)
11. The following hematologic parameters:

    * Hemoglobin > 9 g/dl
    * White blood cell (WBC) > 1000/mm(3)
    * Absolute neutrophil count (ANC) > 750/mm(3)
    * Platelets > 75,000/mm(3)
    * Prothrombin time (PT) and partial thromboplastin time (PTT) less than or equal to 120% of control, unless patient has the presence of a lupus anticoagulant
12. The following hepatic parameters:

    * Bilirubin less than or equal to 1.5 times upper limit of normal (ULN) unless the patient is receiving protease inhibitor therapy (i.e. indinavir, ritonavir, nelfinavir, and atazanavir) known to be associated with increased bilirubin: in this case total bilirubin less than or equal to 7.5 mg/dl and the direct fraction is less than or equal to 0.7 mg/dl.
    * Aspartate aminotransferase (AST)/glutamic oxaloacetic transaminase (GOT) less than or equal to 2.5 times the upper limit of normal
13. Either serum creatinine less than or equal to 1.5 mg/dL or measured creatinine clearance greater than or equal to 60 mL/min
14. Either urine protein <1+ or measured 24 hour urine protein < 500 milligram
15. Able to take aspirin 81mg daily.
16. Study participant must use birth control measure prior to study entry (during screening), during study participation, and for 12 weeks after bevacizumab is discontinued.
17. Inclusion of women and minorities: Both men and women and members of all races and ethnic groups are eligible for this trial.

EXCLUSION CRITERIA:

1. Inability to provide informed consent.
2. KS therapy other than HAART within 3 weeks.
3. History of cumulative doxorubicin or liposomal doxorubicin dose >430 mg/m(2).
4. Supraphysiologic doses of corticosteroids within 3 weeks.
5. Major surgical procedure (including periodontal) within 4 weeks.
6. Surgical or other non-healing wounds, other than KS ulcers.
7. Pregnancy (because of unknown potential for fetal malformation).
8. Breast feeding (because of unknown potential for adverse infant developmental consequences).
9. Has an uncontrolled illness including, but not limited to, ongoing or active infection requiring intravenous (IV) antibiotics, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, cirrhosis, or psychiatric illness/social situations that would limit adherence to study requirements.
10. Past or present history of malignant tumors other than KS unless: a) in a complete remission for greater than or equal to 1 year from the time a response was first documented; b) completely resected basal cell carcinoma; or c) in situ squamous cell carcinoma of the cervix or anus
11. Severe or life-threatening infection within 2 weeks of entry onto the study.
12. History of deep venous or arterial thrombotic disease (including but not limited to, acute myocardial infarction due to coronary thrombosis, ischemic stroke, and peripheral arterial disease), unless:

    * Line-related thrombosis without embolus
    * Occurring greater than or equal to 1 year prior to screening
13. Known procoagulant disorder including prothrombin gene mutation 20210, antithrombin III deficiency, protein c deficiency, protein S deficiency and antiphospholipid syndrome but not including heterozygosity for the Factor V Leiden mutation or the presence of a lupus anticoagulant in the absence of other criteria for the antiphospholipid syndrome.
14. Known bleeding diathesis.
15. History of severe gastrointestinal bleeding within 6 months. Patients with gastrointestinal blood loss due to KS may be included.
16. Hemoptysis within 4 weeks.
17. Substantial central nervous system (CNS) disease including.

    * History of CNS bleeding.
    * Mass lesions in the brain.
    * Uncontrolled seizure disorder.
    * Recent history of cerebrovascular accident (CVA) (e.g. within the past 6 months).
18. Proteinuria > 500 mg/24hrs.
19. Patients with any other abnormality that would be scored as a grade 3 or greater toxicity, except:

    * Lymphopenia
    * Direct manifestations of KS
    * Direct manifestation of HIV
    * Direct manifestation of HIV therapy (i.e. Hyperbilirubinemia associated with protease inhibitors)
    * Asymptomatic hyperuricemia
    * Hypophosphatemia
20. Previous bevacizumab within 6 weeks prior to enrollment.
21. Known hypersensitivity to bevacizumab, Chinese hamster ovary cell products, or other recombinant human or humanized antibodies.
22. Any other condition, including the presence of laboratory abnormalities, which in the opinion of the Principal Investigator or Lead Associate Investigator, places the subject at unacceptable risk if there were to participate in the study or confounds the ability to interpret data from the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-04-23 (Actual); Primary Completion 2015-05-13 (Actual); Study Completion 2017-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Yarchoan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2009-C-0130.html

RESULTS

PARTICIPANT FLOW:
Groups:
- KS; Classic or HIV+ Not Improved on Antivirals: Kaposi's sarcoma (KS) in patients who are Human immunodeficiency virus (HIV) Negative, HIV infected with stable disease for one year despite antiretroviral therapy or progressive disease despite 4 months of antiretroviral therapy.
  Liposomal Doxorubicin: Induction phase dose: Intravenous (IV) bevacizumab 15 mg/kg once, followed 7 days later by liposomal doxorubicin mg/m^2 and bevacizumab every 3 weeks for six cycles.
  Bevacizumab: Induction phase dose: Intravenous (IV) bevacizumab 15 mg/kg once, followed 7 days later by liposomal doxorubicin mg/m^2 and bevacizumab every 3 weeks for six cycles. Maintenance phase dose: IV bevacizumab every 3 weeks for 11 cycles.
- All Other Advanced HIV-associated Kaposi's Sarcoma (KS): All other patients with advanced AIDS-associated KS
  Liposomal Doxorubicin: Induction phase dose: Intravenous (IV) bevacizumab 15 mg/kg once, followed 7 days later by liposomal doxorubicin mg/m^2 and bevacizumab every 3 weeks for six cycles.
  Bevacizumab: Induction phase dose: Intravenous (IV) bevacizumab 15 mg/kg once, followed 7 days later by liposomal doxorubicin mg/m^2 and bevacizumab every 3 weeks for six cycles. Maintenance phase dose: IV bevacizumab every 3 weeks for 11 cycles.
Period: Overall Study
Arm/Group | KS; Classic or HIV+ Not Improved on Antivirals | All Other Advanced HIV-associated Kaposi's Sarcoma (KS)
Started | 10 | 6
Completed | 2 | 3
Not Completed | 8 | 3
Not completed — progressive disease on study | 2 | 1
Not completed — Adverse Event | 2 | 1
Not completed — Lost to follow up | 2 | 0
Not completed — Continuing in follow up period | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KS; Classic or HIV+ Not Improved on Antivirals | All Other Advanced HIV-associated Kaposi's Sarcoma (KS) | Total
Number analyzed (Participants) | 10 | 6 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 6 | 16
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 50.85 [24.8 to 57.1] | 40.85 [32.0 to 57.9] | 45.95 [24.8 to 57.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 6 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 7 | 4 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 4 | 0 | 4
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 10 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) of Six Cycles of Liposomal Doxorubicin Combined With Bevacizumab in Patients With Advanced KS.
Description: Overall response rate is complete response + clinical complete response + partial response. The overall response rate is the fraction of subjects with an overall response after 6 cycles of liposomal doxorubicin in combination with bevacizumab. Response was assessed by a modification of the Acquired Immune Deficiency Syndrome Clinical Trial Group Oncology Committee criteria. Complete response is the absence of any detectable residual disease, including tumor-associated edema, persisting for at least 4 weeks. Clinical complete response is the absence of any detectable residual disease, including tumor associated edema. persisting for at least 4 weeks. Partial response is no progressive disease (increase of 25% or more over baseline in the number of lesions and/or size (sum of the products of the largest perpendicular diameters of the marker lesions) & noting that single lesions which split up into 2 or more smaller lesions during the course of treatment will still be counted as 1.
Time Frame: 6 cycles, an average of 18 weeks
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | KS; Classic or HIV+ Not Improved on Antivirals | All Other Advanced HIV-associated Kaposi's Sarcoma (KS)
Number analyzed (Participants) | 10 | 6
percentage of participants | 50 [27 to 73] | 67 [33 to 91]

2. Secondary Outcome: Complete Response Rate After 6 Cycles of Liposomal Doxorubicin Combined With Bevacizumab
Description: Complete response rate is the fraction of subjects with an complete response after 6 cycles of liposomal doxorubicin in combination with bevacizumab. Response was assessed by a modification of the Acquired Immune Deficiency Syndrome Clinical Trial Group Oncology Committee criteria. Complete response is the absence of any detectable residual disease, including tumor-associated edema, persisting for at least 4 weeks. In patients whom pigmented macular skin lesions persist after apparent complete response, biopsy of at least one representative lesion is required to document the absence of malignant cells. In patients known to have had visceral disease, an attempt at restaging with appropriate endoscopic or radiographic procedures should be made. If such procedures are medically contraindicated, the patient may be classified as having a clinical complete response.
Time Frame: 6 cycles, an average of 18 weeks
Population: No patients had a complete response.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | KS; Classic or HIV+ Not Improved on Antivirals | All Other Advanced HIV-associated Kaposi's Sarcoma (KS)
Number analyzed (Participants) | 10 | 6
percentage of participants | 0 [0 to 21] | 0 [0 to 32]

3. Secondary Outcome: Count of Participants With Serious and Non-serious Adverse Events
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v3.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: 7 years and 6 months and 21 days
Measure: Count of Participants; unit: Participants
Groups:
- KS; Classic or HIV+ Not Improved on Antivirals: Kaposi's sarcoma (KS) in patients who are Human immunodeficiency virus (HIV) Negative, HIV infected with stable disease for one year despite antiretroviral therapy or progressive disease despite 4 months of antiretroviral therapy.
  Liposomal Doxorubicin: Induction phase dose: Intravenous (IV) bevacizumab 15 mg/kg once, followed 7 days later by liposomal doxorubicin mg/m2^ and bevacizumab every 3 weeks for six cycles.
  Bevacizumab: Induction phase dose: Intravenous (IV) bevacizumab 15 mg/kg once, followed 7 days later by liposomal doxorubicin mg/m^2 and bevacizumab every 3 weeks for six cycles. Maintenance phase dose: IV bevacizumab every 3 weeks for 11 cycles.
Arm/Group | KS; Classic or HIV+ Not Improved on Antivirals | All Other Advanced HIV-associated Kaposi's Sarcoma (KS)
Number analyzed (Participants) | 10 | 6
Participants | 10 | 6

4. Secondary Outcome: Median Number of Cycles Need to Obtain a Partial Response
Description: Response was assessed by a modification of the Acquired Immune Deficiency Syndrome Clinical Trial Group Oncology Committee criteria. Partial response is no progressive disease (increase of 25% or more over baseline in the number of lesions and/or size (sum of the products of the largest perpendicular diameters of the marker lesions) and noting that single lesions which split up into 2 or more smaller lesions during the course of treatment will still be counted as 1; no new lesions occurring in previously uninvolved areas of the body; no new visceral sites of involvement or the appearance or worsening of tumor-associated edema or effusions and a 50% or greater decrease in the number and/or size of previously existing lesions lasting for at least 4 weeks or complete flattening of at least 50% of all previously raised lesions (i.e., 50% of all previously nodular or plaque-like lesions become macular) lasting for at least 4 weeks.
Time Frame: 6 cycles, an average of 18 weeks
Measure: Median (95% Confidence Interval); unit: Cycles
Arm/Group | KS; Classic or HIV+ Not Improved on Antivirals | All Other Advanced HIV-associated Kaposi's Sarcoma (KS)
Number analyzed (Participants) | 10 | 6
Cycles | 2 [1 to 6] | 4 [1 to 5]

5. Secondary Outcome: Percentage of Participants With 12- Month Progression-free Survival (PFS)
Description: Participants who survived and were progression free for 12 months. Response was assessed by a modification of the Acquired Immune Deficiency Syndrome Clinical Trial Group Oncology Committee criteria. Progressive disease is an increase of 25% or more over baseline in the number of lesions and/or size (sum of the products of the largest perpendicular diameters) of the marker lesions or a change in character from macular to plaque-like or nodular of at least 25% of the lesions or new visceral sites of involvement or progression of visceral disease or the development of new or increasing tumor-associated edema or effusion that lasts at least 1 week and interfered with the patient's normal activities.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- KS; Classic or HIV+ Not Improved on Antivirals: Kaposi's sarcoma (KS) in patients who are Human immunodeficiency virus (HIV) Negative, HIV infected with stable disease for one year despite antiretroviral therapy or progressive disease despite 4 months of antiretroviral therapy.
  Liposomal Doxorubicin: Induction phase dose: Intravenous (IV) bevacizumab 15 mg/kg once, followed 7 days later by liposomal doxorubicin mg/m^2 and bevacizumab every 3 weeks for six cycles.
  Bevacizumab: Induction phase dose: Intravenous (IV) bevacizumab 15 mg/kg once, followed 7 days later by liposomal doxorubicin mg/m2^ and bevacizumab every 3 weeks for six cycles. Maintenance phase dose: IV bevacizumab every 3 weeks for 11 cycles.
Arm/Group | KS; Classic or HIV+ Not Improved on Antivirals | All Other Advanced HIV-associated Kaposi's Sarcoma (KS)
Number analyzed (Participants) | 10 | 6
percentage of participants | 44 [23 to 64] | 42 [15 to 67]

ADVERSE EVENTS:
Time Frame: 7 years and 6 months and 21 days
Arm/Group | KS; Classic or HIV+ Not Improved on Antivirals | All Other Advanced HIV-associated Kaposi's Sarcoma (KS)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/6
Other Adverse Events (participants affected / at risk) | 10/10 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KS; Classic or HIV+ Not Improved on Antivirals (N=10) | All Other Advanced HIV-associated Kaposi's Sarcoma (KS) (N=6)
Hemorrhage, GI::Rectum (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KS; Classic or HIV+ Not Improved on Antivirals (N=10) | All Other Advanced HIV-associated Kaposi's Sarcoma (KS) (N=6)
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 7 (26) | 5 (17)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 8 (28) | 5 (16)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 4 (12) | 5 (38)
Alkaline phosphatase (Metabolism and nutrition disorders) | 2 (4) | 3 (26)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 (1) | 1 (1)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 2 (2) | 0 (0)
Amylase (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anal bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1 (6) | 2 (26)
CD4 count (Blood and lymphatic system disorders) | 5 (9) | 2 (7)
CNS cerebrovascular ischemia (Nervous system disorders) | 1 (1) | 0 (0)
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 3 (11) | 5 (15)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (1) | 1 (4)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Cholesterol, serum-high (hypercholesteremia) (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Constipation (Gastrointestinal disorders) | 2 (3) | 3 (3)
Constitutional Symptoms - Other (R leg swelling) (General disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 2 (4)
Creatinine (Metabolism and nutrition disorders) | 1 (1) | 2 (10)
Dental: periodontal disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dental: teeth (Gastrointestinal disorders) | 2 (4) | 1 (1)
Dermatology/Skin - Skin breakdown (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Abrasion
Diarrhea (Gastrointestinal disorders) | 2 (3) | 3 (7)
Discoloration of Hard Palate (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (7)
Edema: limb (Blood and lymphatic system disorders) | 4 (8) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 5 (12) | 3 (6)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 (2) | 0 (0)
Flushing (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
GGT (gamma-Glutamyl transpeptidase) (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Gastrointestinal - Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) — Reflux
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 4 (11) | 3 (5)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (1) | 2 (4)
Gum bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 2 (4) | 0 (0)
Hemoglobin (Metabolism and nutrition disorders) | 7 (21) | 5 (29)
Hemoglobinuria (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hemorrhage, GI::Abdomen NOS (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhage, GI::Oral cavity (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hemorrhage, GU::Urinary NOS (Gastrointestinal disorders) | 1 (1) | 3 (6)
Hemorrhage, pulmonary/upper respiratory::Nose (Renal and urinary disorders) | 3 (3) | 4 (17)
Hot flashes/flushes (Endocrine disorders) | 0 (0) | 2 (2)
Hypercholesterolemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hypertension (Cardiac disorders) | 4 (8) | 1 (4)
Dermatology/Skin-Rash:acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — Folliculitis L groin
Infection with normal ANC or Grade 1 or 2 neutrophils::Anal/perianal (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Bronchus (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Colon (Infections and infestations) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Dental-tooth (Infections and infestations) | 2 (2) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils::Oral cavity-gums (gingivitis) (Infections and infestations) | 2 (2) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Upper airway NOS (Infections and infestations) | 4 (5) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils::Urinary tract NOS (Infections and infestations) | 0 (0) | 1 (1)
Infection with unknown ANC::Dental-tooth (Infections and infestations) | 0 (0) | 1 (2)
Infection with unknown ANC::Upper airway NOS (Infections and infestations) | 2 (2) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 6 (35) | 4 (43)
Lymphopenia (Blood and lymphatic system disorders) | 8 (34) | 5 (25)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 2 (2) | 3 (7)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 5 (6) | 2 (2)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Mood alteration::Anxiety (Nervous system disorders) | 1 (2) | 0 (0)
Mood alteration::Depression (Nervous system disorders) | 1 (2) | 0 (0)
Mucositis/stomatitis (clinical exam)::Oral cavity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis/stomatitis (clinical exam)::Stomach (Gastrointestinal disorders) | 1 (2) | 0 (0)
Musculoskeletal/Soft Tissue - Other (Aches/Myalgia; Muscle spasm) (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Nail changes (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal discharge (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (5) | 2 (2)
Neck heaviness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neurology - Other (Burning smell) (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy: sensory (Nervous system disorders) | 4 (4) | 2 (3)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 5 (35) | 4 (42)
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Pain - Right posterior knee (General disorders) | 0 (0) | 1 (1) — 8/10
Pain::Abdomen NOS (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain::Anus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain::Back (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Pain::Bone (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Pain::Extremity-limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain::Head/headache (Nervous system disorders) | 5 (6) | 1 (1)
Pain::Joint (Musculoskeletal and connective tissue disorders) | 4 (5) | 1 (1)
Pain::Muscle (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (2)
Pain::Neck (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain::Oral cavity (Gastrointestinal disorders) | 0 (0) | 1 (2)
Pain::Oral-gums (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain::Pain NOS (General disorders) | 2 (2) | 1 (1)
Pain::Rectum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain::Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Pain::Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Pain::Urethra (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Paresthesia (Nervous system disorders) | 2 (3) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 5 (20) | 3 (3)
Platelets (Blood and lymphatic system disorders) | 6 (21) | 1 (1)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 2 (4) | 2 (2)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Proteinuria (Metabolism and nutrition disorders) | 5 (13) | 3 (18)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Psychosis (hallucinations/delusions) (Nervous system disorders) | 0 (0) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (9)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hemorrhage/Bleeding-Hemorrhage, GU (Renal and urinary disorders) | 0 (0) | 1 (1) — Hematuria
Rhinorrhea (Immune system disorders) | 1 (1) | 0 (0)
Runny nose (Immune system disorders) | 2 (2) | 0 (0)
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 3 (3) | 4 (6)
Sweating (diaphoresis) (General disorders) | 0 (0) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 0 (0) | 1 (1)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1 (1) | 1 (1)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 3 (3) | 1 (1)
Triglyceride, serum-high (hypertriglyceridemia) (Metabolism and nutrition disorders) | 2 (2) | 2 (5)
Ulcer, GI::Anus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ulcer, GI::Rectum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ulceration (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Upper respiratory (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 4 (8) | 1 (6)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dermatology/Skin - Rash: acne/acneform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Folliculitis
Dermatology/Skin - Hand-foot Syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4) — Rash: hand-foot skin reaction
Dermatology/Skin - Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) — Maculo-papular rash; Skin desquamation sole of L foot
Dermatology/Skin - Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Skin discoloration-hands
Dermatology/Skin - Dermal change (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Skin thickening
Metabolic/Laboratory-"Urobilinogen" t (Metabolism and nutrition disorders) | 0 (0) | 1 (4) — Urobilinogen 2-3
Infection - Other, Ungual, foot (Infections and infestations) | 1 (1) | 1 (1) — Fungal foot rash
Musculoskeletal/Soft Tissue, Other-fasciitis, plantar (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Plantar fascilitis
Pulmonary/Upper Respiratory-Nasal cavity/paranasal sinus (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — Sinusitis
Pain - Leg (General disorders) | 0 (0) | 1 (1) — Leg
Pain - Left foot (General disorders) | 1 (1) | 0 (0) — Sole of left foot
Pain - Left middle finger (General disorders) | 0 (0) | 1 (1) — Left middle finger
Pain - Right foot (General disorders) | 1 (1) | 0 (0) — Right foot pain
Pain - Thigh (General disorders) | 1 (1) | 0 (0) — Thigh
Pain - Neck, back, shoulder (General disorders) | 1 (2) | 0 (0) — Neck, back, shoulder pain
Hemorrhage/Bleeding-Hemorrhage, GI (Gastrointestinal disorders) | 1 (1) | 1 (1) — Hematochezia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/36/NCT00923936/Prot_000.pdf
  • Informed Consent Form (2014-06-17): https://cdn.clinicaltrials.gov/large-docs/36/NCT00923936/ICF_001.pdf